CLINICAL TRIAL: NCT00442936
Title: A Multicenter, Double-Blind, Placebo-Controlled, Parallel Group Study to Compare the Response to a Single Treatment With Oral MK0974 With Placebo and Comparator in Subjects With Moderate to Severe Acute Migraine With or Without Aura
Brief Title: Study of Telcagepant (MK-0974) in Participants With Moderate to Severe Acute Migraine With or Without Aura (MK-0974-011)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0974-011; MK-0974-011 (Other: Merck Protocol Number); 2006_525 (Other: Telerx ID Number)
Record Dates: First submitted 2007-02-28; First posted 2007-03-05 (Estimated); Results first posted 2014-08-04 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-09

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — zolmitriptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Telcagepant 150 mg (Experimental): Participants receive telcagepant 150 mg capsules, one capsule administered orally at initial onset of moderate to severe migraine headache. If, after 2 hours post-dose, participants still have a moderate to severe migraine or migraine recurs, participants may receive an optional second dose of study drug (telcagepant 150 mg or placebo) or one dose of non-study rescue medication.
  Interventions: Drug: Telcagepant potassium 150 mg; Drug: Placebo to tecagepant 300 mg; Drug: Placebo to zolmitriptan 5 mg; Drug: Rescue medication
- Telcagepant 300 mg (Experimental): Participants receive telcagepant 300 mg capsules, one capsule administered orally at initial onset of moderate to severe migraine headache. If, after 2 hours post-dose, participants still have a moderate to severe migraine or migraine recurs, participants may receive an optional second dose of study drug (telcagepant 300 mg or placebo) or one dose of non-study rescue medication.
  Interventions: Drug: Telcagepant potassium 300 mg; Drug: Placebo to telcagepant 150 mg; Drug: Placebo to zolmitriptan 5 mg; Drug: Rescue medication
- Zolmitriptan 5 mg (Active Comparator): Participants receive zolmitriptan 5 mg tablets, one tablet administered orally at initial onset of moderate to severe migraine headache. If, after 2 hours post-dose, participants still have a moderate to severe migraine or migraine recurs, participants may receive an optional second dose of study drug (placebo) or one dose of non-study rescue medication.
  Interventions: Drug: Zolmitriptan 5 mg; Drug: Placebo to telcagepant 150 mg; Drug: Placebo to tecagepant 300 mg; Drug: Rescue medication
- Placebo (Placebo Comparator): Participants receive placebo matching capsules or tablets, one capsule or tablet administered orally at initial onset of moderate to severe migraine headache. If, after 2 hours post-dose, participants still have a moderate to severe migraine or migraine recurs, participants may receive an optional second dose of study drug (placebo) or one dose of non-study rescue medication.
  Interventions: Drug: Placebo to telcagepant 150 mg; Drug: Placebo to tecagepant 300 mg; Drug: Placebo to zolmitriptan 5 mg; Drug: Rescue medication

INTERVENTIONS:
Drug: Telcagepant potassium 150 mg — Telcagepant 150 mg liquid-filled soft gel capsules
  Arms: Telcagepant 150 mg
Drug: Telcagepant potassium 300 mg — Telcagepant 300 mg liquid-filled soft gel capsules
  Arms: Telcagepant 300 mg
Drug: Zolmitriptan 5 mg — Zolmitriptan 5 mg tablets
  Arms: Zolmitriptan 5 mg
Drug: Placebo to telcagepant 150 mg — Placebo to match telcagepant 150 mg liquid-filled soft gel capsules
  Arms: Placebo; Telcagepant 300 mg; Zolmitriptan 5 mg
Drug: Placebo to tecagepant 300 mg — Placebo to match tecagepant 300 mg liquid-filled soft gel capsules
  Arms: Placebo; Telcagepant 150 mg; Zolmitriptan 5 mg
Drug: Placebo to zolmitriptan 5 mg — Placebo to match zolmitriptan 5 mg tablets
  Arms: Placebo; Telcagepant 150 mg; Telcagepant 300 mg
Drug: Rescue medication — If moderate or severe migraine headache pain continues or recurs 2 hours after dose of study drug, participants are allowed to take an optional second dose of study drug or their own non-study rescue migraine medication, which may include analgesics (e.g., nonsteroidal anti-inflammatory drugs [NSAIDs] or opiates), anti-emetics, or zolmitriptan. Triptans other than zolmitriptan and ergot derivatives are prohibited for 24 hours following the last dose of study drug.

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of telcagepant (MK-0974) compared to an approved medication for acute migraine. This study was conducted as a "triple-dummy" design; for each dose of study drug, participants each received 3 forms of study drug (2 capsules of active and/or placebo and 1 tablet of active and/or placebo) and were instructed to take one of each form of study drug at dosing time.

The primary hypotheses of this study are that telcagepant is superior to placebo in Pain Freedom at 2 Hours Post-Dose, Pain Relief at 2 Hours Post-Dose, Absence of Photophobia at 2 Hours Post-Dose, Absence of Phonophobia at 2 Hours Post-Dose and Absence of Nausea at 2 Hours Post-Dose.

ELIGIBILITY:
Inclusion Criteria:

* Has at least 1 year history of migraine (with or without aura)
* Females of child bearing potential must use acceptable contraception throughout trial.

Exclusion Criteria:

* Is pregnant/breast-feeding (or is a female expecting to conceive during study period)
* Has history or evidence of stroke/transient ischemic attacks, heart disease, coronary artery vasospasm, other significant underlying cardiovascular diseases, uncontrolled hypertension (high blood pressure), uncontrolled diabetes, or human immunodeficiency virus (HIV) disease
* Has major depression, other pain syndromes that might interfere with study assessments, psychiatric conditions, dementia, or significant neurological disorders (other than migraine)
* Has a history of gastric, or small intestinal surgery, or has a disease that causes malabsorption
* Has a history of cancer within the last 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1380 (Actual)
Dates: Start 2007-02-15 (Actual); Primary Completion 2007-10-02 (Actual); Study Completion 2007-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Ho TW, Ferrari MD, Dodick DW, Galet V, Kost J, Fan X, Leibensperger H, Froman S, Assaid C, Lines C, Koppen H, Winner PK. Efficacy and tolerability of MK-0974 (telcagepant), a new oral antagonist of calcitonin gene-related peptide receptor, compared with zolmitriptan for acute migraine: a randomised, placebo-controlled, parallel-treatment trial. Lancet. 2008 Dec 20;372(9656):2115-23. doi: 10.1016/S0140-6736(08)61626-8. Epub 2008 Nov 25. PMID 19036425
- [Derived] Ho TW, Olesen J, Dodick DW, Kost J, Lines C, Ferrari MD. Antimigraine efficacy of telcagepant based on patient's historical triptan response. Headache. 2011 Jan;51(1):64-72. doi: 10.1111/j.1526-4610.2010.01790.x. Epub 2010 Nov 4. PMID 21054362
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0974-011&kw=0974-011&tab=access

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Telcagepant 150 mg | Telcagepant 300 mg | Zolmitriptan 5 mg | Placebo
Started | 333 | 354 | 345 | 348
Completed | 332 | 354 | 344 | 347
Not Completed | 1 | 0 | 1 | 1
Not completed — Protocol Violation | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telcagepant 150 mg | Telcagepant 300 mg | Zolmitriptan 5 mg | Placebo | Total
Number analyzed (Participants) | 333 | 354 | 345 | 348 | 1380
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.7 (11.2) | 42.6 (11.4) | 41.7 (11.7) | 42.3 (11.6) | 42.3 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 277 | 300 | 298 | 294 | 1169
  Male | 56 | 54 | 47 | 54 | 211

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Pain Freedom (PF) at 2 Hours Post-Dose
Description: Participants were asked to rate their migraine headache severity with ratings of 0=No pain, 1=Mild pain, 2=Moderate pain, and 3=Severe pain. PF at 2 hours post-dose is defined as a decrease from a moderate or severe migraine headache (Grade 2 or 3) at baseline to no pain (Grade 0) at 2 hours post-dose.
Time Frame: 2 hours post-dose
Population: The population consisted of all participants who were randomized, took at least one dose of study drug, recorded a baseline pain score, and had at least one pain score measurement within 2 hours post-dose.
Measure: Number; unit: Participants
Arm/Group | Telcagepant 150 mg | Telcagepant 300 mg | Zolmitriptan 5 mg | Placebo
Number analyzed (Participants) | 317 | 338 | 328 | 328
Participants | 56 | 89 | 101 | 29
Statistical Analysis 1: Comparison: Telcagepant 150 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.26, 95% CI 2-sided [1.40 to 3.66] — From logistic model adjusting for geographic region, baseline migraine severity, and age. An odds ratio >1 is in favor of the first treatment group of the corresponding pairwise comparison
Statistical Analysis 2: Comparison: Telcagepant 300 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.81, 95% CI 2-sided [2.42 to 6.00] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Number of Participants With Pain Relief (PR) at 2 Hours Post-Dose
Description: Participants were asked to rate their migraine headache severity with ratings of 0=No pain, 1=Mild pain, 2=Moderate pain, and 3=Severe pain. PR at 2 hours post-dose is defined as a shift from a moderate or severe migraine headache (Grade 2 or 3) at baseline to mild or no pain (Grade 1 or 0) at 2 hours post-dose.
Time Frame: 2 hours post-dose
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Telcagepant 150 mg | Telcagepant 300 mg | Zolmitriptan 5 mg | Placebo
Number analyzed (Participants) | 317 | 338 | 328 | 328
Participants | 157 | 183 | 185 | 88
Statistical Analysis 1: Comparison: Telcagepant 150 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.82, 95% CI 2-sided [2.02 to 3.95] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Telcagepant 300 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.44, 95% CI 2-sided [2.47 to 4.79] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Number of Participants With Absence of Photophobia at 2 Hours Post-Dose
Description: Participants were asked if they experienced any sensitivity to light. The number of participants who experienced no photophobia (sensitivity to light) at 2 hours post-dose was determined.
Time Frame: 2 hours post-dose
Population: The population consisted of all participants who were randomized, took at least one dose of study drug, recorded a baseline photophobia assessment, and had at least one photophobia assessment within 2 hours post-dose.
Measure: Number; unit: Participants
Arm/Group | Telcagepant 150 mg | Telcagepant 300 mg | Zolmitriptan 5 mg | Placebo
Number analyzed (Participants) | 317 | 338 | 328 | 327
Participants | 143 | 169 | 163 | 92
Statistical Analysis 1: Comparison: Telcagepant 150 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.14, 95% CI 2-sided [1.54 to 2.97] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Telcagepant 300 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.61, 95% CI 2-sided [1.89 to 3.61] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Number of Participants With Absence of Phonophobia at 2 Hours Post-Dose
Description: Participants were asked if they experienced any sensitivity to sound. The number of participants who experienced no phonophobia (sensitivity to sound) at 2 hours post-dose was determined.
Time Frame: 2 hours post-dose
Population: The population consisted of all participants who were randomized, took at least one dose of study drug, recorded a baseline phonophobia assessment, and had at least one phonophobia assessment within 2 hours post-dose.
Measure: Number; unit: Participants
Arm/Group | Telcagepant 150 mg | Telcagepant 300 mg | Zolmitriptan 5 mg | Placebo
Number analyzed (Participants) | 317 | 338 | 326 | 327
Participants | 170 | 193 | 180 | 120
Statistical Analysis 1: Comparison: Telcagepant 150 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.05, 95% CI 2-sided [1.49 to 2.82] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Telcagepant 300 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.37, 95% CI 2-sided [1.73 to 3.25] — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: Number of Participants With Absence of Nausea at 2 Hours Post-Dose
Description: Participants were asked if they experienced any nausea. The number of participants who experienced no nausea at 2 hours post-dose was determined.
Time Frame: 2 hours post-dose
Population: The population consisted of all participants who were randomized, took at least one dose of study drug, recorded a baseline nausea assessment, and had at least one nausea assessment within 2 hours post-dose.
Measure: Number; unit: Participants
Arm/Group | Telcagepant 150 mg | Telcagepant 300 mg | Zolmitriptan 5 mg | Placebo
Number analyzed (Participants) | 316 | 337 | 327 | 327
Participants | 212 | 218 | 232 | 179
Statistical Analysis 1: Comparison: Telcagepant 150 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.73, 95% CI 2-sided [1.25 to 2.39] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Telcagepant 300 mg vs Placebo; Test type: Superiority or Other; p = 0.006, Regression, Logistic; Odds Ratio (OR) = 1.55, 95% CI 2-sided [1.13 to 2.13] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Number of Participants With Sustained Pain Freedom (SPF) From 2 to 24 Hours Post-Dose
Description: SPF is defined as PF at 2 hours post-dose with no return of mild/moderate/severe headache through 24 hours post-dose, and with no administration of either the optional second dose of study drug or any rescue medication between 2 and 24 hours post-dose.
Time Frame: 2 to 24 hours post-dose
Population: The population consisted of all participants who were randomized, took at least one dose of study drug, recorded a baseline pain score, had at least one pain score measurement within 2 hours post-dose, and had at least one pain score measurement at between 2 and 24 hours post-dose.
Measure: Number; unit: Participants
Arm/Group | Telcagepant 150 mg | Telcagepant 300 mg | Zolmitriptan 5 mg | Placebo
Number analyzed (Participants) | 314 | 336 | 328 | 328
Participants | 34 | 66 | 59 | 14
Statistical Analysis 1: Comparison: Telcagepant 150 mg vs Placebo; Test type: Superiority or Other; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 2.80, 95% CI 2-sided [1.47 to 5.35] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Telcagepant 300 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 5.75, 95% CI 2-sided [3.15 to 10.51] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Number of Participants With Total Migraine Freedom (TMF) at 2 Hours Post-Dose
Description: TMF at 2 hours post-dose is defined as PF at 2 hours post-dose without any of the following migraine-related symptoms: phonophobia, photophobia, nausea or vomiting at 2 hours post-dose.
Time Frame: 2 hours post-dose
Population: The population consisted of all participants who were randomized, took at least one dose of study drug, recorded a baseline pain score, had at least one pain score measurement within 2 hours post-dose, and had at least one assessment for phonophobia, photophobia, nausea and vomiting within 2 hours post-dose.
Measure: Number; unit: Participants
Arm/Group | Telcagepant 150 mg | Telcagepant 300 mg | Zolmitriptan 5 mg | Placebo
Number analyzed (Participants) | 317 | 338 | 328 | 328
Participants | 43 | 76 | 87 | 27
Statistical Analysis 1: Comparison: Telcagepant 150 mg vs Placebo; Test type: Superiority or Other; p = 0.026, Regression, Logistic; Odds Ratio (OR) = 1.78, 95% CI 2-sided [1.07 to 2.97] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Telcagepant 300 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.34, 95% CI 2-sided [2.08 to 5.35] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Number of Participants With Total Migraine Freedom (TMF) at 2 to 24 Hours Post-Dose
Description: TMF at 2 to 24 hours post-dose is defined as TMF at 2 hours post-dose with no administration of either the optional second dose of study drug or any rescue medication between 2 and 24 hours post-dose, no return of mild/moderate/severe headache within 24 hours and no presence of phonophobia, photophobia, nausea or vomiting within 24 hours post-dose.
Time Frame: 2 to 24 hours post-dose
Population: The population consisted of all participants who were randomized, took at least one dose of study drug, recorded a baseline pain score, had at least one pain score measurement within 2 to 24 hours post-dose, and had at least one assessment for phonophobia, photophobia, nausea and vomiting within 2 to 24 hours post-dose.
Measure: Number; unit: Participants
Arm/Group | Telcagepant 150 mg | Telcagepant 300 mg | Zolmitriptan 5 mg | Placebo
Number analyzed (Participants) | 315 | 336 | 328 | 328
Participants | 26 | 57 | 51 | 13
Statistical Analysis 1: Comparison: Telcagepant 150 mg vs Placebo; Test type: Superiority or Other; p = 0.021, Regression, Logistic; Odds Ratio (OR) = 2.25, 95% CI 2-sided [1.13 to 4.47] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Telcagepant 300 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 5.21, 95% CI 2-sided [2.78 to 9.76] — [estimate comment as in outcome 1, analysis 1]

9. Primary Outcome: Number of Participants Who Experience At Least One Adverse Event (AE)
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the product. Participants were monitored for occurrence AEs for up to 14 days after last dose study drug. Participants who took both active and placebo study drug were counted in the active group.
Time Frame: Up to 14 days after last dose of study drug
Population: The population consisted of all participants who received at least one dose of study drug. Participants were included in the treatment arm corresponding to the study treatment actually taken at the time of the AE.
Measure: Number; unit: Participants
Arm/Group | Telcagepant 150 mg | Telcagepant 300 mg | Zolmitriptan 5 mg | Placebo
Number analyzed (Participants) | 334 | 352 | 345 | 349
Participants | 105 | 131 | 175 | 112

10. Primary Outcome: Number of Participants Who Discontinue Study Drug Due to an AE
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the product. Participants who took both active and placebo study drug were counted in the active group.
Time Frame: Up to 48 hours after first dose of study drug
Population: The populaton consisted of all participants who received at least one dose of study drug. Participants were included in the treatment arm corresponding to the study treatment actually taken at the time of the AE.
Measure: Number; unit: Participants
Arm/Group | Telcagepant 150 mg | Telcagepant 300 mg | Zolmitriptan 5 mg | Placebo
Number analyzed (Participants) | 334 | 352 | 345 | 349
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 14 days after last dose of study drug
Description: The All Participants as Treated population consisted of all participants who received at least 1 dose of study drug. Participants were included in the treatment arm corresponding to the study treatment actually taken at the time of the AE.
Arm/Group | Telcagepant 150 mg | Telcagepant 300 mg | Zolmitriptan 5 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/334 | 0/352 | 0/345 | 1/349
Other Adverse Events (participants affected / at risk) | 66/334 | 74/352 | 107/345 | 54/349
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telcagepant 150 mg (N=334) | Telcagepant 300 mg (N=352) | Zolmitriptan 5 mg (N=345) | Placebo (N=349)
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Telcagepant 150 mg (N=334) | Telcagepant 300 mg (N=352) | Zolmitriptan 5 mg (N=345) | Placebo (N=349)
Dry mouth (Gastrointestinal disorders) | 18 | 21 | 28 | 13
Nausea (Gastrointestinal disorders) | 13 | 17 | 20 | 13
Fatigue (General disorders) | 14 | 15 | 24 | 8
Dizziness (Nervous system disorders) | 15 | 19 | 38 | 20
Paraesthesia (Nervous system disorders) | 4 | 6 | 18 | 5
Somnolence (Nervous system disorders) | 15 | 19 | 20 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation.